CLINICAL TRIAL: NCT02602600
Title: Effect of Glucagon-like Peptide-1 Stimulation on Coronary Microvascular Dysfunction in Women With Angina Pectoris and no Obstructive Stenosis of Major Coronary Vessels
Brief Title: Glucagon-like Peptide-1 and Coronary Microvascular Dysfunction in Women With Angina Pectoris and no Coronary Stenosis
Acronym: GAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eva Prescott (Other)
Responsible Party: Sponsor-Investigator, Eva Prescott, MD, DMSc, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAP
Record Dates: First submitted 2015-11-08; First posted 2015-11-11 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Microvascular Angina
MeSH Terms: conditions — Microvascular Angina | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Liraglutide (Experimental): Liraglutide up to 3.0 mg daily injected subcutaneously (minimum 1.2 mg daily) for 12 weeks followed by 2 weeks of weight maintenance diet. Before initiating treatment participants will serve as their own controls for 4 weeks.
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: Liraglutide — * Liraglutide up to 3 mg daily injected subcutaneously (minimum 1.2 mg daily) for 12 weeks.
  * Weight maintenance diet for 2 weeks
  Other Names: Victoza

SUMMARY:
The aim of the present study is to evaluate the effect of treatment with Liraglutide on the coronary microvasculature and angina symptoms, in overweight patients with microvascular dysfunction and angina pectoris but no coronary artery stenosis.

DETAILED DESCRIPTION:
Background:

Patients with symptoms and signs of ischemia are referred to coronary angiography (CAG) or CT angiography (CT-CAG). A significant proportion of these patients and especially women appear to have no obstructive coronary stenosis. Patients with angina-like symptoms and no macrovascular coronary stenosis have previously been considered without increased risk of major cardiovascular events, but novel data indicate that this assumption may not be true.

Abnormal coronary flow and metabolic response to stress have been reported, which is consistent with a possible microvascular ethology for the symptoms. Both endothelium- and non-endothelium dependent impaired coronary reactivity may contribute. The endothelium dependent component has been linked to risk factors and pro-inflammatory processes promoting atherosclerosis. The non-endothelium dependent mechanisms may involve vascular smooth muscle cells, undergoing alterations in phenotype in response to physiological and pathophysiological stimuli like hypertension and diabetes.

Both invasive and non-invasive diagnostic methods are available for the assessment of coronary microvascular dysfunction. In the absence of a flow limiting stenosis upstream, indirect measurement is possible by using transthoracic Doppler stress echocardiography (TTDSE). TTDSE provides assessment of coronary blood flow velocity in one of the major coronary vessels that can be used to determine coronary flow velocity reserve (CFR) after hyperemia. This method does primarily assess the non-endothelium dependent component of coronary microvascular dysfunction.

Despite reassurance that no stenosis on major coronary vessels is found, many patients continue to have chest pain resulting in emergency visits, hospitalizations and repeat cardiac catheterizations with adverse effect on quality of life, employment and health care costs.

Treatment options for patients with angina symptoms are lacking when no macrovascular coronary stenosis is found. Standard anti-angina treatments are usually tried, but do not relieve symptoms in many of these patients.

Preclinical studies with Glucagon-like peptide-1 (GLP-1) and GLP-1 receptor (GLP-1R) agonists demonstrate cardioprotective effects. However, the underlying mechanisms are often not well defined. Many studies do not distinguish between direct versus indirect actions of GLP-1R agonists, nor take into account the potential actions of the cleavage product, GLP-1. GLP-1R is found in atrial cardiomyocytes in animal models and in the sinoatrial node in humans. Furthermore endothelial cells and vascular smooth muscle cells seem to be targets for GLP-1 action. In animal models GLP-1 promotes myocardial glucose uptake independent of insulin, increases contractility and coronary flow and improves outcome and survival after myocardial infarction in vivo. Limited data exists on the cardioprotective effect of GLP-1 in humans. A few studies have evaluated the effect of GLP-1 in patients presenting acute myocardial infarction or stenosis of major coronary vessels, whereas no data exists on the effect in patients with stable coronary artery disease. Two randomized studies have investigated the effect of GLP-1 infusion in ST-elevation acute myocardial infarction, and found reduced infarct size at three months follow-up. Several small pilot studies in patients with coronary heart disease have found that GLP-1 infusion or dipeptidyl peptidase-4 inhibitor improves left ventricular ejection fraction. None of the human trials have involved prolonged treatment with GLP-1.

Data from previous work suggest that GLP-1 and weight loss may have beneficial effects on microvascular circulation and cardiovascular risk factors. In a small cross-over study of 20 patients with type2 diabetes but no angina, 10 weeks of GLP1-R agonist treatment (Liraglutide, 1,2 mg/day) led to a small but insignificant improvement in coronary microcirculation, concomitant with a significant decrease in body weight and blood pressure and improvement in glycemic control. Another study included overweight patients with ischemic heart disease and found, that a mean weight loss of 10.6% achieved through a low energy diet improved microvascular function (CFR) and coronary risk factors such as blood pressure, lipid profile, and glycemic control (non-diabetics) as well as symptoms. Thus data on any cardioprotective effect of long-term treatment with GLP-1 in humans is sparse, and it may be speculated that any beneficial effect may be due to the weight lowering effect.

Objective The aim of the present study is to evaluate the effect of treatment with Liraglutide on the coronary microvasculature and angina symptoms, in overweight patients with microvascular dysfunction (CFR≤2,5) and angina pectoris but no coronary artery stenosis.

Hypothesis Liraglutide improves microvascular function and alleviates symptoms in women with angina pectoris and microvascular coronary dysfunction, but no obstructive stenosis of major coronary vessels.

Design An open label trial consisting of a four-weeks control period without intervention, followed by Liraglutide 3 mg once daily for 12 weeks + 2 weeks of weight maintenance diet. Study participants will serve as their own controls during the first four weeks not receiving treatment. Outcome parameters will be measured at baseline and at 4 and 18 weeks. The first two measurements (baseline and four weeks measurements) will in this way serve as documentation of the variance of repeated measurements. Blinding of participants and investigators will not be possible due to the study setup, but investigators will be blinded to pre- and posttreatment measurements when analysing results at the end of the study. Furthermore investigator will be blinded to previous CFR measurements during data collection.

Study drug Liraglutide s a once daily human GLP-1 analogue with 97% linear amino-acid sequence homology to human GLP-1. Liraglutide works by stimulating the release of insulin only when glucose levels become too high and by inhibiting appetite. It lowers blood glucose with the unique advantage that glucose lowering ceases when blood glucose gets into the normal range. Liraglutide is approved in the EU and US for the treatment of type 2 diabetes mellitus at doses up to 1,8 mg administered subcutaneously once daily. Recently the US Food and Drug Administration (FDA) and the European Medicines Agency (EMA) have approved Liraglutide as obesity treatment. The indication is as an adjunct to lifestyle modifications for chronic weight management in individuals with a body mass index (BMI) of ≥30 kg/m2, or BMI≥27 kg/m2 with at least one weight-related comorbidity such as dysglycaemia (pre-diabetes or type 2 diabetes mellitus), hypertension, dyslipidaemia or obstructive sleep apnoea. The max dose for obesity treatment is 3.0 mg daily.

When prescribed with the aim of weight loss, Liraglutide is administrated subcutaneously and titrated up to the maximally recommended dosage for obesity. By treating participants on the indication overweight interference with other antihyperglycemic medications is avoided. Treatment is initiated with 0.6 mg once daily for one week and increased weekly until the recommended max dose of 3 mg. If it is not possible to reach maximal dosage due to adverse effects, the participants will stay at the highest dose tolerated. Participants will be excluded if they do not tolerate a treatment dose of at least 1.2 mg Liraglutide per day, since a lower dosage is unlikely to result in a weight loss of at least 5% .Treatment duration will be 12 weeks and the last two weeks will consist of a weight maintenance diet before outcome measurements are done. On this dosage and duration a weight loss of at least 5% is expected. Participants will be advised to reduce calorie intake and increase physical activity. Control of compliance will be made at visits by telephone calls (structured open questions interviews) Furthermore participants will note every time the medication is taken in a diary.

Participants Study participants will be recruited from an ongoing multicenter study of women with symptoms and signs of angina pectoris, 'Improving diagnosis and treatment of women with angina pectoris and microvascular disease (iPower)'. Before inclusion in the iPower study, participants have undergone CAG or CT-CAG with no significant stenosis of major coronary vessels. As part of the iPower study the coronary flow reserve is measured by transthoracic doppler stress echocardiography with dipyridamole induces stress.

Diagnostic methods Fasting blood samples will be collected. Some of the blood samples will be stored in a biobank. Blood samples will be stored until the end of the study (last patient, last visit) plus five years, and the blood samples will be destroyed thereafter.

Angina symptoms will be assess by the Seattle Angina Questionnaire (SAQ) which is a 19-item health-related quality-of-life measure for patients with coronary artery disease.

A score change of 10 points is clinically perceptible to patients and is considered a clinically relevant difference, while a substantial change is considered to be a change of 20 points.

Echocardiographic measurements of CFR, systolic and diastolic function including strain will be done both at rest and during dipyridamole induced stress. CFR is calculated as the ratio between coronary flow velocity during hyperemia and rest. Coronary microvascular dysfunction is defined as CFR<2.5.

Endothelial function will be measured by flow mediated dilation (FMD). Peripheral endothelial function correlates well with coronary endothelial function.

A whole body dual X-ray absorptiometry (DEXA) scan will be performed at baseline and after 18 weeks to estimate body composition.

Statistics There are two main outcomes: Microvascular function assessed by CFR and symptom burden assessed by SAQ.

CFR is a continuous response variable. A difference in repeated measurements within each subject is found to be normally distributed with a standard deviation 0.35. If the mean change in CFR post treatment is 0.23, the investigators will need to study 27 subjects to be able to reject the null hypothesis that there will be no change in the mean CFR with probability (power) 0.9. The Type I error probability associated with this test of the null hypothesis is 0.05. At least 33 participants will be included in anticipation of around 20% drop-out.

SAQ has four subscales each with a score from 1-100. According to previous studies a change in SAQ score of 10 points is perceptible by the patients and therefore clinically meaningful. The investigators have not found data on within-study subject variation on SAQ. However, previous trials have obtained changes in SAQ of 10-20 points after an intervention. Based on these findings the investigators expect to see a change in SAQ score of at least 10 point. By estimating a SD of 15, it is calculated that 26 study subjects is sufficient to attain a statistical power of >90% to detect a significant difference of 10 points post treatment in any SAQ item.

For the remaining secondary outcomes, if the response is normally distributed, the investigators will be able to detect a true difference in the mean response of participants of 0.66 x the SD of the within group change with a probability (power) 0.9. The Type I error probability associated with this test of the null hypothesis, that the population mean is unchanged after the intervention, is 0.05.

Monitoring:

The study will be monitored by the unit for Good Clinical Practice (GCP-unit) at the University of Copenhagen. Quality checks of data, data registry procedures and source data verification will be performed by the GCP-unit.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 40-75 with angina-like symptoms assessed by the Seattle Angina Questionnaire (SAQ).
* Women aged 40-75 with angina-like symptoms assessed by the Seattle Angina Questionnaire (SAQ).
* Referred for ischemic heart disease (IHD) assessment with no significant coronary stenosis (>50%) at coronary angiography or CT-angiography
* Impaired CFR assessed by echo Doppler flow (defined ratio≤2,5).
* BMI≥25kg/m2

Exclusion Criteria:

* Allergy to dipyridamole, theophyllamine or liraglutide
* Previous myocardial infarction or revascularization
* No episodes of chest pain within 6 months before inclusion
* Diabetes (reported, noted in journal or patient on antidiabetic medication)
* Other causes of chest discomfort deemed highly likely
* Left ventricular ejection fraction <45
* Significant valvular disease
* Congenital heart disease
* severe co-morbidity with limited life-expectancy< 1 year
* Severe asthma
* Severe chronic obstructive pulmonary disease
* Pregnancy (pregnancy test will be done at inclusion)
* No use of contraception although in child-bearing age. A woman is regarded fertile, following menarche and until becoming post-menopausal unless permanently sterile. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. The birth control methods considered safe and effective includes combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), intrauterine device (IUD) and intrauterine hormone-releasing system ( IUS). Women in child-bearing age will have to use one of the above mentioned contraceptive methods from inclusion in the study until the end of study participation.
* physical or mental disability
* active cancer
* significant renal (eGRF<30) or hepatic co-morbidity
* chronic alcohol abuse
* atrial fibrillation
* Atrio-ventricular block>1st degree
* chronic or previous acute pancreatitis
* inflammatory bowel disease
* history of thyroid carcinoma
* participation in other clinical trial if relevant for the present study.
* Language- or other barrier to giving informed consent
* No signed informed consent

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-11-19 (Actual); Primary Completion 2017-04-18 (Actual); Study Completion 2017-04-18 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Coronary Flow Reserve | Assessed at baseline, week 4 and week 18
  Assessed by transthoracic doppler stress echocardiography
Change from baseline in Angina Symptoms | Assessed at baseline, week 4 and week 18
  Assessed by the Seattle Angina Questionnaire

SECONDARY OUTCOMES:
Change in endothelial function | Assessed at baseline, week 4 and week 18
  Assessed by Flow Mediated Dilation of the brachial artery by ultrasound
Change in cardiac function | Assessed at baseline, week 4 and week 18
  Assessed by speckle tracking echocardiography
Change in body weight | Assessed at baseline, week 4 and week 18
Change in body composition | Assessed before and after treatment (week 4 and week 18)
  Assessed by dexa scan

CONTACTS AND LOCATIONS:
Overall Officials: Eva IB Prescott, MD, DMSc, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg University Hospital, Copenhagen, Copenhagen Northwest, Denmark

REFERENCES:
- [Result] Patel MR, Peterson ED, Dai D, Brennan JM, Redberg RF, Anderson HV, Brindis RG, Douglas PS. Low diagnostic yield of elective coronary angiography. N Engl J Med. 2010 Mar 11;362(10):886-95. doi: 10.1056/NEJMoa0907272. PMID 20220183
- [Result] Jespersen L, Hvelplund A, Abildstrom SZ, Pedersen F, Galatius S, Madsen JK, Jorgensen E, Kelbaek H, Prescott E. Stable angina pectoris with no obstructive coronary artery disease is associated with increased risks of major adverse cardiovascular events. Eur Heart J. 2012 Mar;33(6):734-44. doi: 10.1093/eurheartj/ehr331. Epub 2011 Sep 11. PMID 21911339
- [Result] Johnson BD, Shaw LJ, Pepine CJ, Reis SE, Kelsey SF, Sopko G, Rogers WJ, Mankad S, Sharaf BL, Bittner V, Bairey Merz CN. Persistent chest pain predicts cardiovascular events in women without obstructive coronary artery disease: results from the NIH-NHLBI-sponsored Women's Ischaemia Syndrome Evaluation (WISE) study. Eur Heart J. 2006 Jun;27(12):1408-15. doi: 10.1093/eurheartj/ehl040. Epub 2006 May 23. PMID 16720691
- [Result] Gulati M, Cooper-DeHoff RM, McClure C, Johnson BD, Shaw LJ, Handberg EM, Zineh I, Kelsey SF, Arnsdorf MF, Black HR, Pepine CJ, Merz CN. Adverse cardiovascular outcomes in women with nonobstructive coronary artery disease: a report from the Women's Ischemia Syndrome Evaluation Study and the St James Women Take Heart Project. Arch Intern Med. 2009 May 11;169(9):843-50. doi: 10.1001/archinternmed.2009.50. PMID 19433695
- [Result] Pepine CJ, Anderson RD, Sharaf BL, Reis SE, Smith KM, Handberg EM, Johnson BD, Sopko G, Bairey Merz CN. Coronary microvascular reactivity to adenosine predicts adverse outcome in women evaluated for suspected ischemia results from the National Heart, Lung and Blood Institute WISE (Women's Ischemia Syndrome Evaluation) study. J Am Coll Cardiol. 2010 Jun 22;55(25):2825-32. doi: 10.1016/j.jacc.2010.01.054. PMID 20579539
- [Result] Reis SE, Holubkov R, Conrad Smith AJ, Kelsey SF, Sharaf BL, Reichek N, Rogers WJ, Merz CN, Sopko G, Pepine CJ; WISE Investigators. Coronary microvascular dysfunction is highly prevalent in women with chest pain in the absence of coronary artery disease: results from the NHLBI WISE study. Am Heart J. 2001 May;141(5):735-41. doi: 10.1067/mhj.2001.114198. PMID 11320360
- [Result] Camici PG, Crea F. Coronary microvascular dysfunction. N Engl J Med. 2007 Feb 22;356(8):830-40. doi: 10.1056/NEJMra061889. No abstract available. PMID 17314342
- [Result] Jespersen L, Abildstrom SZ, Hvelplund A, Madsen JK, Galatius S, Pedersen F, Hojberg S, Prescott E. Burden of hospital admission and repeat angiography in angina pectoris patients with and without coronary artery disease: a registry-based cohort study. PLoS One. 2014 Apr 4;9(4):e93170. doi: 10.1371/journal.pone.0093170. eCollection 2014. PMID 24705387
- [Result] Di Franco A, Villano A, Di Monaco A, Lamendola P, Russo G, Stazi A, Scavone G, Nerla R, Sestito A, Lanza GA, Crea F. Correlation between coronary microvascular function and angina status in patients with stable microvascular angina. Eur Rev Med Pharmacol Sci. 2014;18(3):374-9. PMID 24563437
- [Result] Ussher JR, Drucker DJ. Cardiovascular actions of incretin-based therapies. Circ Res. 2014 May 23;114(11):1788-803. doi: 10.1161/CIRCRESAHA.114.301958. PMID 24855202
- [Result] Nikolaidis LA, Elahi D, Hentosz T, Doverspike A, Huerbin R, Zourelias L, Stolarski C, Shen YT, Shannon RP. Recombinant glucagon-like peptide-1 increases myocardial glucose uptake and improves left ventricular performance in conscious dogs with pacing-induced dilated cardiomyopathy. Circulation. 2004 Aug 24;110(8):955-61. doi: 10.1161/01.CIR.0000139339.85840.DD. Epub 2004 Aug 16. PMID 15313949
- [Result] Ban K, Noyan-Ashraf MH, Hoefer J, Bolz SS, Drucker DJ, Husain M. Cardioprotective and vasodilatory actions of glucagon-like peptide 1 receptor are mediated through both glucagon-like peptide 1 receptor-dependent and -independent pathways. Circulation. 2008 May 6;117(18):2340-50. doi: 10.1161/CIRCULATIONAHA.107.739938. Epub 2008 Apr 21. PMID 18427132
- [Result] Noyan-Ashraf MH, Momen MA, Ban K, Sadi AM, Zhou YQ, Riazi AM, Baggio LL, Henkelman RM, Husain M, Drucker DJ. GLP-1R agonist liraglutide activates cytoprotective pathways and improves outcomes after experimental myocardial infarction in mice. Diabetes. 2009 Apr;58(4):975-83. doi: 10.2337/db08-1193. Epub 2009 Jan 16. PMID 19151200
- [Result] Lonborg J, Kelbaek H, Vejlstrup N, Botker HE, Kim WY, Holmvang L, Jorgensen E, Helqvist S, Saunamaki K, Terkelsen CJ, Schoos MM, Kober L, Clemmensen P, Treiman M, Engstrom T. Exenatide reduces final infarct size in patients with ST-segment-elevation myocardial infarction and short-duration of ischemia. Circ Cardiovasc Interv. 2012 Apr;5(2):288-95. doi: 10.1161/CIRCINTERVENTIONS.112.968388. Epub 2012 Apr 10. PMID 22496084
- [Result] Woo JS, Kim W, Ha SJ, Kim JB, Kim SJ, Kim WS, Seon HJ, Kim KS. Cardioprotective effects of exenatide in patients with ST-segment-elevation myocardial infarction undergoing primary percutaneous coronary intervention: results of exenatide myocardial protection in revascularization study. Arterioscler Thromb Vasc Biol. 2013 Sep;33(9):2252-60. doi: 10.1161/ATVBAHA.113.301586. Epub 2013 Jul 18. PMID 23868944
- [Result] McCormick LM, Kydd AC, Read PA, Ring LS, Bond SJ, Hoole SP, Dutka DP. Chronic dipeptidyl peptidase-4 inhibition with sitagliptin is associated with sustained protection against ischemic left ventricular dysfunction in a pilot study of patients with type 2 diabetes mellitus and coronary artery disease. Circ Cardiovasc Imaging. 2014 Mar;7(2):274-81. doi: 10.1161/CIRCIMAGING.113.000785. Epub 2014 Feb 6. PMID 24503784
- [Result] Read PA, Khan FZ, Heck PM, Hoole SP, Dutka DP. DPP-4 inhibition by sitagliptin improves the myocardial response to dobutamine stress and mitigates stunning in a pilot study of patients with coronary artery disease. Circ Cardiovasc Imaging. 2010 Mar;3(2):195-201. doi: 10.1161/CIRCIMAGING.109.899377. Epub 2010 Jan 14. PMID 20075143
- [Result] Read PA, Hoole SP, White PA, Khan FZ, O'Sullivan M, West NE, Dutka DP. A pilot study to assess whether glucagon-like peptide-1 protects the heart from ischemic dysfunction and attenuates stunning after coronary balloon occlusion in humans. Circ Cardiovasc Interv. 2011 Jun;4(3):266-72. doi: 10.1161/CIRCINTERVENTIONS.110.960476. Epub 2011 May 17. PMID 21586690
- [Result] Read PA, Khan FZ, Dutka DP. Cardioprotection against ischaemia induced by dobutamine stress using glucagon-like peptide-1 in patients with coronary artery disease. Heart. 2012 Mar;98(5):408-13. doi: 10.1136/hrt.2010.219345. Epub 2011 May 10. PMID 21561896
- [Result] Nikolaidis LA, Mankad S, Sokos GG, Miske G, Shah A, Elahi D, Shannon RP. Effects of glucagon-like peptide-1 in patients with acute myocardial infarction and left ventricular dysfunction after successful reperfusion. Circulation. 2004 Mar 2;109(8):962-5. doi: 10.1161/01.CIR.0000120505.91348.58. Epub 2004 Feb 23. PMID 14981009
- [Result] Faber R, Zander M, Pena A, Michelsen MM, Mygind ND, Prescott E. Effect of the glucagon-like peptide-1 analogue liraglutide on coronary microvascular function in patients with type 2 diabetes - a randomized, single-blinded, cross-over pilot study. Cardiovasc Diabetol. 2015 Apr 22;14:41. doi: 10.1186/s12933-015-0206-3. PMID 25896352
- [Result] Pedersen LR, Olsen RH, Jurs A, Astrup A, Chabanova E, Simonsen L, Wisloff U, Haugaard SB, Prescott E. A randomised trial comparing weight loss with aerobic exercise in overweight individuals with coronary artery disease: The CUT-IT trial. Eur J Prev Cardiol. 2015 Aug;22(8):1009-17. doi: 10.1177/2047487314545280. Epub 2014 Jul 31. PMID 25082954
- [Derived] Suhrs HE, Raft KF, Bove K, Madsbad S, Holst JJ, Zander M, Prescott E. Effect of liraglutide on body weight and microvascular function in non-diabetic overweight women with coronary microvascular dysfunction. Int J Cardiol. 2019 May 15;283:28-34. doi: 10.1016/j.ijcard.2018.12.005. Epub 2019 Jan 2. PMID 30773266